CLINICAL TRIAL: NCT01871714
Title: Phenotypic Properties in Individuals Affected With X-linked Hypohidrotic Ectodermal Dysplasia: Symptoms and Facial Recognition
Brief Title: Phenotypic Properties in Individuals Affected With XLHED
Acronym: ECP-014
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-014
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: X Linked Hypohidrotic Ectodermal Dysplasia
Keywords: XLHED; HED; Hypohidrotic Ectodermal Dysplasia; X Linked Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Genetic tests will be carried out in a subset of subject in order to confirm XLHED status.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- XLHED affected Males: All males ages 4 and up affected by XLHED
- Females affected by XLHED: Adult females (ages 18-45) affected by XLHED
- Unaffected females: Unaffected adult female controls (ages 18-45)

SUMMARY:
The current study design incorporates two previously developed, non-invasive approaches to characterize the phenotype of individuals affected with XLHED.

DETAILED DESCRIPTION:
The current study design incorporates two previously developed, non-invasive approaches to characterize the phenotype of individuals affected with XLHED. Facial 3-dimensional (3D) imaging will be created from white-field morphometric scanning (Hammond, 2004. The 3D facial photographs collected from males (ages 4 years and up) will be used to develop a non-invasive screening tool, which could enable detection of craniofacial signs of XLHED in the newborn period. 3D facial profiling has been reported to be effective in identifying HED (Dellavia et al., 2008), but the technology does not yet meet the ease-of-use criteria for a universal screening tool.

Standard 2-dimensional (2D) frontal and lateral facial photographs will be taken of the same XLHED-affected male subjects as well as of adult females (ages 18-45 yrs) at risk for being XLHED carriers and unaffected adult female controls. The 2D facial photographs will serve a dual purpose; the first being to beta-test a previously developed algorithm to identify males affected with XLHED (Automatic Phenotype Identification of XLHED Patients Final Report, December 25, 2012, unpublished), and the second to adapt the facial recognition algorithm to identify female carriers of XLHED.

ELIGIBILITY:
Inclusion Criteria:

1. Females of original gender of age 18-45 years who are registered and attending the 2013 NFED Family Conference. This will include those at risk for XLHED and controls
2. XLHED-affected males of original gender of age 4 yrs and up who are registered and attending the 2013 NFED Family Conference
3. Provide informed consent/assent

Exclusion Criteria:

1. Subjects who are not able or are not willing to comply with the procedures of this protocol
2. Subjects with any major medical problem that will prevent them from participating in this study
3. Male subjects who participated in the prior study ECP-003 sponsored by Edimer Pharmaceuticals Inc. in May 2011 in San Francisco, CA
4. Males at risk for XLHED with prior genetic testing that did not reveal an EDA mutation

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: XLHED affected males and females and unaffected female controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To collect demographic and clinical status information in XLHED-affected males, adult females at risk for XLHED and adult female controls | Study day 1
  To collect demographic and clinical status information in XLHED-affected males, adult females at risk for XLHED and adult female controls using a medical questionnaire
To test and refine a computer algorithm for facial recognition of XLHED | Study day 1
  To test and refine a computer algorithm for facial recognition of XLHED based on 2D facial photographs obtained from subjects at risk for XLHED and controls
To evaluate 3-dimensional facial imaging technology for mapping craniofacial development in XLHED males | Study day 1
  To evaluate 3-dimensional facial imaging technology for mapping craniofacial development in XLHED males
To test for the presence of genetic mutations in subjects at risk for XLHED | Study day 1
  To test for the presence of genetic mutations in subjects at risk for XLHED who lack prior genetic diagnosis
To test the validity of a using saliva samples for genetic testing | Study day 1
  To test the validity of a using saliva samples for genetic testing buy simultaneously perform genetic testing on blood and salvia and comparing the mutations identified

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Omni Houston Hotel, Houston, Texas, United States

REFERENCES:
- See also: Sponsor website — http://edimerpharma.com